CLINICAL TRIAL: NCT04316546
Title: A Multi-Cohort Phase 2 Dose-Escalation Study of MK-7075 (Miransertib) in Proteus Syndrome
Brief Title: MK-7075 (Miransertib) in Proteus Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200034; 20-HG-0034
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12-17

CONDITIONS: Proteus Syndrome
Keywords: AKT1; CCTN; Mosaic Overgrowth Disorder
MeSH Terms: conditions — Proteus Syndrome | interventions — Miransertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-7075 (miransertib) (Experimental): This is a single-arm study. All study participants will be taking the experimental drug, MK-7075 (miransertib).
  Interventions: Drug: MK-7075 (miransertib)

INTERVENTIONS:
Drug: MK-7075 (miransertib) — MK-7075 (miransertib) is a small molecule developed by ArQule Inc., a wholly owned subsidiary of Merck Sharp & Dohme (Merck), that effectively inhibits AKT. Proteus syndrome is caused by mosaic activating mutations in AKT1. This is a Phase 2 trial investigating the efficacy of miransertib as a treatment for adult and pediatric patients with Proteus syndrome.

SUMMARY:
Background:

Proteus syndrome is a rare overgrowth disorder. Most people begin to have symptoms between 6 months and 2 years of age. There are very few living adults with this disease. There is also no known treatment for it. Researchers want to see if a new drug can slow down or stop overgrowth in people with Proteus syndrome.

Objective:

To learn if miransertib is a safe and effective treatment for Proteus syndrome.

Eligibility:

People ages 3 and older with Proteus syndrome.

Design:

Participants will be screened with a medical checkup. They will answer questions about their medical history and current health. They will have a physical exam with vital signs. They will have an electrocardiogram to measure their heartbeat. They will give blood and urine samples. They will repeat the screening tests during the study.

Participants will take a miransertib pill once a day. They will bring their empty pill bottles with them to the NIH when they visit. If they can t swallow a pill, researchers will try to find other ways for them to take the drug.

Participants will have X-rays, ultrasounds, and imaging scans. Photos may be taken of their feet and other parts of the body that have or develop signs of Proteus syndrome.

Participants will have lung function tests to measure how much and how fast air moves out of their lungs.

Participants will complete surveys about their levels of pain, physical functioning, and quality of life.

Participants may have additional tests performed to assess their individual disease. They may have consultations with other specialists.

Participation lasts about 4 years. Participants will have 20-30 visits at the NIH.

DETAILED DESCRIPTION:
Study Description: The primary objective of this study is to determine the response rate of miransertib as measured by the change in cerebriform connective tissue nevus (CCTN) involvement of the plantar surface from baseline, using blinded independent central review of lesional photography in individuals with Proteus syndrome (Cohort 1). Cohorts 2 and 3 will enroll additional patients whose non-plantar CCTN Proteus syndrome-associated lesions will be evaluated to address the secondary and exploratory study objectives. All participants will be treated with miransertib in continuous, 28-day cycles. Participants in Cohorts 1 and 2 will receive miransertib at the starting dose of 15 mg/m^2 daily for the first three cycles, and then the dose will be increased to 25 mg/m^2 daily, provided no clinically significant drug-related toxicity is observed. Participants in Cohort 3 will receive miransertib at the dose they were on at the time of enrollment if continuing use of miransertib or at the starting dose for Cohorts 1 and 2, not to exceed 45 mg/dose daily. Safety and toxicity data will be gathered on all participants. Participants will stay on treatment for up to 52 cycles. The final clinical safety follow-up will be performed 30 days after the last dose.

Objectives:

Primary Objective: To determine the response to treatment with miransertib as measured by the growth of plantar CCTN in individuals with Proteus syndrome.

Secondary Objectives:

1. To estimate the change from baseline in pain in participants treated with miransertib
2. To estimate change from baseline in physical functioning in participants treated with miransertib
3. To estimate change from baseline in quality of life in participants treated with miransertib
4. To describe the long-term tolerability and safety of miransertib
5. To determine the duration of response in responders with respect to the primary study endpoint

Exploratory Objectives:

1. To describe the effect of miransertib on Proteus syndrome-related overgrowth manifestations.
2. To describe the effect of miransertib on the rate of growth of the CCTN lesion as compared to historical data from untreated participants
3. To determine if the clinical gestalt status of participants with Proteus syndrome improves on/after treatment with miransertib
4. To describe the effect of miransertib on D-dimer and fibrinogen levels
5. To describe the PK profile of miransertib

Endpoints:

Primary Endpoint (assessed in Cohort 1):

Change in lesion proportion of the plantar surface will be used to classify each participant as either a responder or non-responder (binary) in the treated population. The primary endpoint is the response rate (defined as a <= 5% increase in the proportion of plantar involvement from baseline after 26 cycles) as assessed by blinded central photography review.

Secondary Endpoints:

1. Change from baseline in pain score as assessed by the NRS-11 Pain Rating Scale
2. Change from baseline in physical functioning as assessed by PROMIS (Pediatric Upper Extremity Short Form 8a, Parent Proxy Upper Extremity Short Form 8a, Pediatric Mobility Short Form 8a, Parent Proxy Mobility Short Form 8a, Physical Function Short Form 8b, Parent Proxy Pain Behavior Short Form 8a)
3. Change from baseline in quality of life as assessed by the Pediatric Quality of Life Inventory (PedsQL)
4. Safety and tolerability as assessed by frequency, duration and severity of AEs from the first dose of miransertib through 30

   days after the last dose of the drug (severity of AEs will be assessed by CTCAE version 5.0)
5. Time from response to failure to respond defined as having a > 5% increase in the proportion of plantar involvement over a 26 cycle period assessed every 6-7 cycles

Exploratory Endpoints:

1. Change from baseline in selected disease-related manifestations, such as those evaluated by imaging (e.g., x-ray, CT, MRI, ultrasound, photography) and/or physical function assessments (e.g., pulmonary function test, six-minute walk test, pegboard test)
2. Behavior of the CCTN lesion while on continuous treatment with miransertib using historical control data for comparison
3. Change in clinical gestalt status in treated participants using a blinded review panel
4. Change from baseline in D-dimer and fibrinogen levels
5. PK parameters (e.g., maximum plasma drug concentration [Cmax], time to maximum plasma drug concentration [Tmax], and area under the curve [AUC]) which are calculated from plasma concentration-time data

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants in all Cohorts must meet the criteria below:

* Signed informed consent, and when applicable, signed assent
* Have a molecular diagnosis of Proteus syndrome with documented somatic AKT1 mutation from a CLIA-certified laboratory or international equivalent.
* Have progressive and measurable disease (e.g., a measurable manifestation of Proteus syndrome with evidence or report of worsening of manifestation(s)/ in the last 12 months)
* Adequate organ function as indicated by the following laboratory values:

Hematological:

* Hemoglobin (Hgb): >=10.0 g/dL
* Glycated hemoglobin (HbA1c): <=8% (<=64 mmol/mol)
* Absolute neutrophil count (ANC): >=1.5 x 10^9/L
* Platelet count >=150 x 10^9/L

Hepatic:

1. Total bilirubin <=2 x upper limit of normal (ULN)
2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=3 x ULN

Renal:

1. Serum creatinine depending on age:

   2-5 years male and female: <=0.50 mg/dL

   6-10 years male and female: <=0.59 mg/dL

   11-15 years male and female: <=1.2 mg/dL

   >15 years male and female: <=1.5 mg/dL

   Metabolic (lipids):
   * Cholesterol: <=400 mg/dL (<=10.34 mmol/L)
   * Triglyceride: <=500 mg/dL (<=5.7 mmol/L)
   * If a female is of child-bearing potential, documentation of a negative pregnancy test is required prior to enrollment. Sexually active participants (male and female) must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse while on study and for up to 90 days after ending treatment
   * Ability to complete the questionnaires by the participant and/or his/her caregiver

   The following specific criteria will be used to assign participants to Cohorts:

   Cohort 1 (Proteus syndrome with plantar CCTN) specific criteria:

   -Have at least one plantar CCTN that can accurately be measured by standardized photography. The CCTN is defined as a nevus with at least two gyri and three sulci affecting 10% - 70% of the total surface area of the foot.

   -Male or female participants age greater than or equal to 3 and less than or equal to 17 years old and BSA of greater than or equal to 0.33 m^2

   Cohort 2 (Proteus syndrome without plantar CCTN) specific criteria:
   * Individuals without an evaluable plantar CCTN
   * No prior exposure to miransertib
   * Male or female participants age >=3 years old and BSA of >=0.33 m^2

   Cohort 3 (Proteus syndrome previously treated with miransertib) specific criteria:

   -Participants previously treated with miransertib or currently receiving miransertib under Compassionate Use/Expanded Access or an existing trial (i.e., 16-HG-0014)

   -Male or female participants greater than or equal to 3 years old BSA of greater than or equal to 0.33 m^2

   Note: All participants must meet Cohort-related age criteria by/on the date of the first dose, Cycle 1 Day 1

   EXCLUSION CRITERIA:

   An individual who meets any of the following criteria will be excluded from participation in this study:

   - History of Type 1 or Type 2 uncontrolled diabetes mellitus requiring regular medication (other than metformin or other oral hypoglycemic agents) or fasting glucose greater than or equal to 160 mg/dL ( if >12 years old) and greater than or equal to 180 mg/dL (if less than or equal to 12 years old) at the baseline/screening visit

   -History of clinically significant cardiac disorders:

   --Myocardial infarction (MI) or congestive heart failure defined as Class II-IV per the New York Heart Association (NYHA) classification within six months of the first dose of miransertib (MI occurring >6 months of the first dose of miransertib will be permitted)

   --Grade 2 (per National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE v 5.0]) or worse conduction defect (e.g., right or left bundle branch block).

   -Major surgery, radiotherapy, chemotherapy, or immunotherapy within four weeks of the first dose of miransertib
   * Any experimental systemic therapy for the purpose of treating Proteus syndrome (e.g., sirolimus, everolimus, high dose steroids, alpelisib) within two weeks of the first dose of miransertib, except for participants who were previously or are currently treated with miransertib under a Compassionate Use/Expanded Access program or existing protocol

     * Participants who were previously treated with or currently are receiving miransertib will be enrolled on Cohort 3 and treated according to the Schedule of Assessments/Study Visits defined in this protocol
   * Intolerance of, or severe toxicity attributed to, AKT inhibitors (e.g., miransertib, uprosertib, afuresertib, ipatasertib)
   * Concurrent severe uncontrolled illness not related to Proteus syndrome

     * Ongoing or active infection
     * Known human immunodeficiency virus (HIV) infection malabsorption syndrome
     * Psychiatric illness/substance abuse/social situation that would limit compliance with study requirements
   * Pregnant or breastfeeding (contraception requirements can be found above and in the informed consent form)
   * Inability to comply with study evaluations or to follow drug administration guidelines
   * Concomitant use of a prohibited medication
   * Regular tobacco use and/or use of cannabidiol/tetrahydrocannabidiol (CBD/THC), and/or vaping products

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
CCTN | Baseline, two years
  Change in CCTN involvement of the plantar surface from baseline will be used to classify each subject as either a responder or non-responder (binary) in the treated population. The primary endpoint is response rate (defined as =< 5% increase in plantar involvement from baseline over 26 cycles). This will be assessed by blinded central photography review.

SECONDARY OUTCOMES:
Quality of life | Periodically throughout the study (described in schedule of activities)
  Change from baseline in pain score (NRS-11), physical functioning (PROMIS), and quality of life (PedsQL).
Long-term safety and tolerability | Periodically throughout the study (described in schedule of activities)
  Periodic safety (e.g., physical examination, vital sign measurements, clinical laboratory tests, use of concomitant medications and collection of AE information) assessments.
Duration of response | Periodically throughout the study (described in schedule of activities)
  Duration of response is defined as the amount of time from first response signal to progression of CCTN involvement >5% over a 26 cycle period assessed every 6-7 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Leslie G Biesecker, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindhurst MJ, Yourick MR, Yu Y, Savage RE, Ferrari D, Biesecker LG. Repression of AKT signaling by ARQ 092 in cells and tissues from patients with Proteus syndrome. Sci Rep. 2015 Dec 11;5:17162. doi: 10.1038/srep17162. PMID 26657992
- [Background] Keppler-Noreuil KM, Sapp JC, Lindhurst MJ, Darling TN, Burton-Akright J, Bagheri M, Dombi E, Gruber A, Jarosinski PF, Martin S, Nathan N, Paul SM, Savage RE, Wolters PL, Schwartz B, Widemann BC, Biesecker LG. Pharmacodynamic Study of Miransertib in Individuals with Proteus Syndrome. Am J Hum Genet. 2019 Mar 7;104(3):484-491. doi: 10.1016/j.ajhg.2019.01.015. Epub 2019 Feb 22. PMID 30803705
- [Background] Nathan NR, Patel R, Crenshaw MM, Lindhurst MJ, Olsen C, Biesecker LG, Keppler-Noreuil KM, Darling TN. Pathogenetic insights from quantification of the cerebriform connective tissue nevus in Proteus syndrome. J Am Acad Dermatol. 2018 Apr;78(4):725-732. doi: 10.1016/j.jaad.2017.10.018. Epub 2017 Oct 16. PMID 29042227
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-HG-0034.html